CLINICAL TRIAL: NCT04832867
Title: Pulmonary Rehabilitation in COVID-19 Patients: The Initial Results of Acute and Subacute Rehabilitation
Brief Title: Pulmonary Rehabilitation in COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Meltem Vural, principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: Pulmonary rehabilitation
Record Dates: First submitted 2021-03-27; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It was aimed to evaluate the respiratory functions of patients who were given respiratory rehabilitation, bed positioning and early mobilization, and the time of leaving the hospital.

DETAILED DESCRIPTION:
According to the clinical classification of the World Health Organization, COVID-19; It manifests itself in a wide spectrum, ranging from mild illness, Pneumonia, Severe pneumonia, Acute respiratory distress syndrome (ARDS), to Sepsis and septic shock, resulting in death. In the presence of acute respiratory failure, a decrease in lung compliance leads to increased respiratory work, impaired blood oxygenation, and rapid and superficial breathing patterns. In this case, minimizing inspiratory effort and maximizing the mechanical efficiency of breathing is the most important approach of treatment. In these clinical conditions, the strength of the respiratory muscles may also be reduced.

The challenge of COVID-19 requires a multidisciplinary approach. Rehabilitative intervention should be a part of the treatment pathway from the early stages of the disease. There is an urgent need to build information based on the most effective non-pharmacological measures to ensure the earliest discharge and best recovery after complex COVID-19 infection. Multimodal rehabilitation at all stages of the disease should be part of a holistic medical approach, but there is still no consensus on the timing and type of intervention.

According to the clinical classification of COVID-19 disease, especially according to the WHO clinical classification, 2.-4. The respiratory system is significantly affected during the stages. In addition, after the active phase of the disease, it is not clear how much damage or sequelae will remain in patients, as there is not enough information about the long-term consequences. In the appropriate patient, pulmonary rehabilitation interventions at the appropriate time will definitely be required.

The aims of pulmonary rehabilitation in general are:

• To keep the respiratory tract open; To reduce respiratory tract resistance and improve ventilation by preventing secretion accumulation with positioning, mobilization, effective cough and other secretion drainage methods, The diaphragm and other respiratory muscles in a more normal position and function.

to ensure that With a breathing pattern that improves the respiratory task and reduces air entrapment reducing the respiratory rate,

* To reduce respiratory work / burden and energy consumption during breathing with appropriate training,
* To prevent or increase chest mobility with exercises suitable for the individual, to detect postural deformities in the musculoskeletal system due to lung disorders, to prevent and / or correct deformity development with appropriate exercise prescription,
* To reduce dyspnea and to relax,
* To improve endurance and general exercise tolerance,
* Suppressing anxiety, depression and anxiety,
* To improve the loss of function and quality of life.

Pulmonary rehabilitation consists of the following items in scope:

Exercise training; respiratory and physical exercise training and breathing strategies

* Work and occupation therapy
* Patient education and smoking cessation
* Nutritional assessment and support
* Psychosocial support
* Long-term oxygen therapy
* Use of non-invasive and invasive mechanical ventilation

Exercise training in pulmonary rehabilitation; It is the most important and obligatory one among the PR elements, it can be thought that it will be the most effective in meeting the PR objectives.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Those who have been hospitalized since 11.01.2020
* Those who have been consulted to the physical therapy clinic since 11.01.2020

Exclusion Criteria:

* Fever ˃38.0 °
* Initial consultation time ˂7 days
* In those with 3 days from the onset of the disease to shortness of breath Chest radiographic scans showing 50% progression within 24 to 48 hours
* With Spo2 level ≤95%
* Resting blood pressure ˂90 / 60 (1mmHg = 0.133kPa) or ˃140 / 90mmHg. 100 heart rate per minute Those with moderate and / or severe heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients in Hospital's service
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
GLASKOW COMA SCALE | change from baseline glaskow coma scale at 1 months
  The scale was described in 1974 by Graham tesdale and Bryan Jenett as a way to communicate of patients with an acute brain injury. A person's GCS score can range from 3 (completely unresponsive) to 15 (responsive). This score is used to guide immediate medical care after a brain injury (such as a car accident) and also to monitor hospitalized patients and track their level of consciousness.
  The glasgow coma scale is often used to help define the severity of TBI. Mild head injuries are generally defined as those associated with a glasgow coma scale score of 13-15, and moderate head injuries are those associated with a glasgow coma scale score of 9-12. A glasgow coma scale score of 8 or less defines a severe head injury.
mMRC dyspnea scale | change from baseline at 1 month
  THe mMRC dsypnea scale quantifies disability attributable to breathlessness and is useful for charecterizing baseline dyspnea in patients with respiratory disease. describes baseline dyspnea but does not accurately quantify response to treatment of chornic obstructive pulmonary disease (COPD).

SECONDARY OUTCOMES:
SpO2 | change from baseline at 1 month
  Oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin (unsaturated + saturated) in the blood. The human body requires and regulates a very precise and specific balance of oxygen in the blood. Normal arterial blood oxygen saturation levels in humans are 95-100 percent.
carbon dioxide (CO2) | change from baseline at 1 month
  The normal range for CO2 is 23 to 29 mEq/L (milliequivalent units per liter of blood). The blood test often measures blood pH along with CO2 levels to further determine the cause of your symptoms. Blood pH is a measurement of acidity or alkalinity.
cardiac output test | change from baseline at 1 month
  Cardiac output (CO), also known as heart output denoted by the symbols {\displaystyle Q}Q, or {\displaystyle {\dot {Q}}_{c}}{\dot Q}_{{c}},[2] is a term used in cardiac physiology that describes the volume of blood being pumped by the heart, by the left and right ventricle, per unit time. Cardiac output (CO) is the product of the heart rate (HR), i.e. the number of heartbeats per minute (bpm), and the stroke volume (SV), which is the volume of blood pumped from the ventricle per beat; thus, CO = HR × SV.[3] Values for cardiac output are usually denoted as L/min. For a healthy person weighing 70 kg, the cardiac output at rest averages about 5 L/min; assuming a heart rate of 70 beats/min, the stroke volume would be approximately 70 ml.

CONTACTS AND LOCATIONS:
Overall Officials: meltem vural, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkor Dr. Sadi Konuk Research and Training hospital, Istanbul, Turkey (Türkiye)